CLINICAL TRIAL: NCT00429767
Title: Reducing Cocaine/Heroin Abuse With SR-Amphetamine and Buprenorphine: Study 1
Brief Title: Sustained Release d-Amphetamine & Buprenorphine on Drug Seeking Behavior in Opioid & Cocaine Dependent Individuals
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NIDA - 022243; R01DA022243 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders; Cocaine Abuse or Dependence
Keywords: Opioid; Cocaine; Drug Self Administration
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether maintenance on different oral doses of sustained release d-amphetamine (SR-AMP) combined with constant-dose sublingual buprenorphine (BUP) is safe and well tolerated and decreases self-administration of cocaine alone or combined with hydromorphone (HYD). Secondary aims are to determine whether SR-AMP attenuates the subjective and physiological effects of cocaine during drug sampling periods prior to choice opportunities.

DETAILED DESCRIPTION:
Heroin abusers also frequently abuse cocaine, and concurrent use of these drugs is associated with more severe drug dependence and associated psychiatric and medical problems, greater risk for HIV infection, worse drug abuse treatment outcome, and creates a public health burden. New methods and solutions are needed for this problem.

While human laboratory models exist to study choice of cocaine or opioids individually, studies have not examined choice of cocaine alone or cocaine/opioid combinations by heroin dependent individuals, nor have there been interventions to reduce such drug use. We recently developed a sensitive laboratory-based choice progressive ratio procedure to study drug-seeking behavior for opioids. This study will extend this procedure, in the form of drug combination vs. money choices, to obtain a novel human laboratory model of cocaine/opioid abuse. The purpose of this study is to determine whether maintenance on different doses of sustained release d-amphetamine (SR-AMP) combined with constant-dose buprenorphine (BUP) is safe and well tolerated and decreases self-administration of cocaine alone or combined with HYD. Secondary aims are to determine whether SR-AMP attenuates the subjective and physiological effects of cocaine during drug sampling periods prior to choice opportunities.

One goal of this new study is to develop a human laboratory model of polydrug abuse by allowing participants (who abuse both heroin and cocaine) to choose between drug combinations or money. The second goal of this study is to develop medication treatments to reduce cocaine use by opioid dependent individuals.

Participants in this observational study will take part in multiple trials in which they have the opportunity to choose between drug combinations (cocaine alone or combined with HYD; relative to HYD alone and dual placebo) or money. On the morning of each session, prior to the choice procedure, participants will receive a sample of the drug dose that can be chosen. Participants will be asked to attend to the effects produced by the drug combination because they will be able to choose this relative to money in the choice task in the afternoon session. During the choice procedure, participants will have 12 opportunities to choose either drug or money. Participants will use a computer to earn choices. Respiration rate, oxygen saturation, heart rate, and blood pressure will be monitored throughout the study. Self-report questionnaires will be completed at different times during the study. Participants will be maintained on a constant dose of BUP throughout the study, with a minimum 2-week lead before the experiment, and a fixed 3-week detoxification after study completion. During the experiment they will be maintained on different doses of SR-AMP and on a constant dose of BUP.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent and Cocaine abuse or dependence, as determined by structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates and cocaine
* Willing to use an adequate form of contraception for the duration of the study
* Reads and writes English

Exclusion Criteria:

* Psychiatric illness, as determined by the DSM-IV criteria
* History of, or current neurological disease, including structural abnormalities, seizures, infectious disease, history of other neurological diseases or head trauma.
* History of cardiovascular disease, myocardial infarction, chest pain or palpations on exertion or drug use
* Systolic blood pressure greater than 160 or less than 95 mmHg; Diastolic blood pressure >95 mmHg
* Clinically abnormal ECG
* Pulmonary disease, including asthma, obstructive pulmonary disease, cor pulmonale, tuberculosis
* Systemic disease (e.g., endocrinopathies, liver or kidney failure, myxedema, hypothyroidism, Addison's disease, autoimmune disease)
* Current alcohol or sedative drug dependence
* Pregnant or breastfeeding
* Currently receiving treatment for a Substance Abuse/Dependence Disorder or seeking treatment
* Been in a research study within the last 30 days
* Known phobia of injections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Heroin dependent and Cocaine abuse or dependent research volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964
- [Derived] Greenwald MK, Lundahl LH, Steinmiller CL. Sustained release d-amphetamine reduces cocaine but not 'speedball'-seeking in buprenorphine-maintained volunteers: a test of dual-agonist pharmacotherapy for cocaine/heroin polydrug abusers. Neuropsychopharmacology. 2010 Dec;35(13):2624-37. doi: 10.1038/npp.2010.175. Epub 2010 Sep 29. PMID 20881947